CLINICAL TRIAL: NCT01958580
Title: A Pilot Safety and Toxicity Trial of Adjuvant Chemotherapy With Gemcitabine and Docetaxel and Radiation Therapy for Completely Resected Uterine Leiomyosarcoma
Brief Title: Gemcitabine Hydrochloride, Docetaxel, and Radiation Therapy in Treating Patients With Uterine Sarcoma That Has Been Removed By Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to low accrual. PI left the institution
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-03-096; NCI-2013-01364 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13-014; 13-03-096 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH)
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Results first posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-07

CONDITIONS: Stage IA Uterine Sarcoma; Stage IB Uterine Sarcoma; Stage IC Uterine Sarcoma; Stage IIA Uterine Sarcoma; Stage IIB Uterine Sarcoma; Stage IIIA Uterine Sarcoma; Stage IIIB Uterine Sarcoma; Stage IIIC Uterine Sarcoma; Stage IVA Uterine Sarcoma; Stage IVB Uterine Sarcoma; Uterine Corpus Leiomyosarcoma
MeSH Terms: interventions — Gemcitabine; Docetaxel; Brachytherapy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (gemcitabine, docetaxel, brachytherapy/IMRT, EBRT) (Experimental): CHEMOTHERAPY: Patients receive gemcitabine hydrochloride IV over 90 minutes on days 1 and 8 and docetaxel IV over 1 hour on day 8. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  RADIATION THERAPY: Beginning week 10, patients undergo 3 fractions of brachytherapy or IMRT over 3 weeks. Patients then undergo EBRT QD 5 days a week for 5 weeks.
  Interventions: Drug: Gemcitabine Hydrochloride; Drug: Docetaxel; Radiation: Internal Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Radiation: External Beam Radiation Therapy; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: Difluorodeoxycytidine (dFdC); dFdCyd
Drug: Docetaxel — Given IV
  Other Names: TXT
Radiation: Internal Radiation Therapy — Undergo brachytherapy
  Other Names: Brachytherapy; Internal Radiation; Internal Radiation Brachytherapy; Radiation Brachytherapy
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam RT
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies gemcitabine hydrochloride, docetaxel, and radiation therapy in treating patients with uterine sarcoma that has been removed by surgery. Drugs used in chemotherapy, such as gemcitabine hydrochloride and docetaxel, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high energy x rays to kill tumor cells. Giving combination chemotherapy with radiation therapy may kill any tumor cells that remain after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the toxicity and tolerability of adjuvant pelvic radiation in combination with gemcitabine (gemcitabine hydrochloride)/docetaxel chemotherapy in patients with stage 1 and 2 surgically-resected uterine leiomyosarcoma.

SECONDARY OBJECTIVES:

I. To assess the two year recurrence-free survival in patients with uterine leiomyosarcoma treated with chemotherapy and radiation therapy including defining the patterns of recurrence in patients with uterine leiomyosarcoma who were treated with this regimen.

OUTLINE:

CHEMOTHERAPY: Patients receive gemcitabine hydrochloride intravenously (IV) over 90 minutes on days 1 and 8 and docetaxel IV over 1 hour on day 8. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

RADIATION THERAPY: Beginning week 10, patients undergo 3 fractions of brachytherapy or intensity modulated radiation therapy (IMRT) over 3 weeks. Patients then undergo external beam radiation therapy (EBRT) once daily (QD) 5 days a week for 5 weeks.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented uterine leiomyosarcoma with no visible residual disease
* Surgical staging to include total hysterectomy, +/- removal of ovaries and fallopian tubes, +/- lymph node sampling
* Patients must be entered no more than 12 weeks post operatively
* Eastern Cooperative Oncology Group (ECOG) performance status of < 2
* Written voluntary informed consent

Exclusion Criteria:

* Serum glutamic oxaloacetic transaminase (SGOT) and /or serum glutamate pyruvate transaminase (SGPT) > 2.5 times the institutional upper limit of normal
* Total serum bilirubin > 1.5 mg/dl
* History of chronic or active hepatitis
* Serum creatinine > 2.0 mg/dl
* Platelets < 100,000/mm3
* Absolute neutrophil count (ANC) < 1500/mm3
* Hemoglobin < 8.0 g/dl (the patient may be transfused prior to study entry)
* Patients with severe or uncontrolled concurrent medical disease (eg. uncontrolled diabetes, unstable angina, myocardial infarction within 6 months, congestive heart failure, etc.)
* Patients with any prior chemotherapy or radiotherapy for pelvic malignancy
* Patients who have had prior therapy with gemcitabine or docetaxel
* Patients with known hypersensitivity to gemcitabine or docetaxel
* Patients with known hypersensitivity to pegfilgrastim and filgrastim
* Patients with any history of cancer with the exception of non-melanoma skin cancer are excluded if there is any evidence of other malignancy being present within the past five years
* Patients with dementia or altered mental status that would prohibit the giving and understanding of informed consent at the time of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-09-17 (Actual); Primary Completion 2017-02-24 (Actual); Study Completion 2017-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akiva Novetsky, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three participants were enrolled into the study between 9/17/2013 and 6/17/2014.
Groups:
- Treatment (Gemcitabine, Docetaxel, Brachytherapy/IMRT/EBRT): CHEMOTHERAPY: Patients receive gemcitabine hydrochloride IV over 90 minutes on days 1 and 8 and docetaxel IV over 1 hour on day 8. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  RADIATION THERAPY: Beginning week 10, patients undergo 3 fractions of brachytherapy or IMRT over 3 weeks. Patients then undergo EBRT QD 5 days a week for 5 weeks.
  Gemcitabine Hydrochloride: Given IV
  Docetaxel: Given IV
  Internal Radiation Therapy: Undergo brachytherapy
  Intensity-Modulated Radiation Therapy: Undergo IMRT
  External Beam Radiation Therapy: Undergo EBRT
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Gemcitabine, Docetaxel, Brachytherapy/IMRT/EBRT)
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Gemcitabine, Docetaxel, Brachytherapy/IMRT, EBRT): CHEMOTHERAPY: Patients receive gemcitabine hydrochloride IV over 90 minutes on days 1 and 8 and docetaxel IV over 1 hour on day 8. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  RADIATION THERAPY: Beginning week 10, patients undergo 3 fractions of brachytherapy or IMRT over 3 weeks. Patients then undergo EBRT QD 5 days a week for 5 weeks.
  Gemcitabine Hydrochloride: Given IV
  Docetaxel: Given IV
  Internal Radiation Therapy: Undergo brachytherapy
  Intensity-Modulated Radiation Therapy: Undergo IMRT
  External Beam Radiation Therapy: Undergo EBRT
  Laboratory Biomarker Analysis: Correlative studies
Arm/Group | Treatment (Gemcitabine, Docetaxel, Brachytherapy/IMRT, EBRT)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants] — Population: patients were lost to followup and were not analyzed
  Participants
    <=18 years | 0
    Between 18 and 65 years | 3
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-free Survival
Description: Two-year recurrence-free survival probability will be estimated, with 95% confidence limits based on exact methods for the binomial distribution. In the event of censoring before two years, a Kaplan-Meier estimate of the survival probability will be used and a Kaplan-Meier survival curve will be estimated and presented as well. The study was terminated prior to analyses
Time Frame: Date of entry to date of reappearance of disease, assessed at 2 years. The study was terminated prior to analyses
Population: Data pertaining to Recurrence-free Survival was not collected/aggregated and therefore not analyzed.
Arm/Group | Treatment (Gemcitabine, Docetaxel, Brachytherapy/IMRT, EBRT)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 1 year following completion of treatment (~69 weeks total)
Arm/Group | Treatment (Gemcitabine, Docetaxel, Brachytherapy/IMRT, EBRT)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Gemcitabine, Docetaxel, Brachytherapy/IMRT, EBRT) (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (2) — Grade 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Gemcitabine, Docetaxel, Brachytherapy/IMRT, EBRT) (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (6) — Episodic. Grade 1-2
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 1
Edema Limbs (General disorders) | 1 (2) — Grade 1-2. Bilateral lower extremities
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) — Grade 1
Nephrotoxicity (Renal and urinary disorders) | 1 (1) — Grade 1
Diarrhea (Gastrointestinal disorders) | 1 (1) — Grade 1
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 1
Peripheral Neuropathy (Nervous system disorders) | 1 (1) — Grade 1
Fatigue (General disorders) | 1 (1) — Grade 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-09): https://cdn.clinicaltrials.gov/large-docs/80/NCT01958580/Prot_SAP_000.pdf